CLINICAL TRIAL: NCT01821807
Title: Postdural Puncture Headache After Spinal Anesthesia for Cesarean Section, Two Different Needles.
Brief Title: Comparison of Two Spinal Needles Regarding Postdural Puncture Headache
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Dr, Adiyaman University Research Hospital
Other Study IDs: PDPH 26Q26A
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural, Headache; Complications; Anesthesia, Spinal and Epidural, in Pregnancy
Keywords: spinal anesthesia; spinal needle; cesarean section; headache; backache
MeSH Terms: conditions — Headache; Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 26 gauge quincke: Patients (n=150) will be treated with 26 gauge quincke spinal needle for spinal anesthesia for cesarean section.
- 26 gauge atraucan: Patients (n=110) will be treated with 26 gauge atraucan spinal needle for spinal anesthesia for cesarean section.

SUMMARY:
The aim of the study is to observe the rate of postdural puncture headache observed after spinal anesthesia in cesarean section patients.

Two kind of spinal anesthesia needles will be used:

1. 26 Gauge Quincke (cutting-tip needle)
2. 26 Gauge Atraucan (atraumatic needle)

The investigators will observe:

1. Number of spinal punctures
2. Time required for the spinal anesthesia procedure

Patients will be evaluated after 7 days for:

1. Headache
2. Backache

DETAILED DESCRIPTION:
It is a known phenomenon that spinal anesthesia sometimes results in headache.

The aim of the study is to observe the rate of postdural puncture headache observed after spinal anesthesia in cesarean section patients.

Two kind of spinal anesthesia needles will be used:

1. 26 Gauge Quincke (cutting-tip needle)
2. 26 Gauge Atraucan (atraumatic needle)

We will observe:

1. Number of spinal punctures
2. Time required for the spinal anesthesia procedure

Patients will be evaluated after 7 days for:

1. Headache
2. Backache

2 kind of spinal anesthesia needles will be used, but no comparison will be made. This is an observational study. Although literature gives different rates of postdural puncture headache for these two needles, we observe the same rate of headache in our clinical practice. We want to define the real rate of postdural puncture headache in patients undergoing cesarean section with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female patients between 18-40 years old undergoing cesarean section
* Patient accepting spinal anesthesia

Exclusion Criteria:

* Infection at the spinal needle insertion cite
* Coagulability disorder
* Patient not accepting the procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant female patients between 18-40 years old undergoing cesarean section in Adiyaman University Research Hospital, Turkey.
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Adiyaman University Research Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the patients in the first month of study were selected in group "Quincke". All the others recruited in the second month of the study were enrolled in group "Atraucan".
Pre-assignment Details: Non-compliance to the suggestions of the investigators for the part of patients and loss of the contact with the patient were criteria for exclusion.
Period: Overall Study
Arm/Group | 26 Gauge Quincke | 26 Gauge Atraucan
Started | 150 | 110
Completed | 147 | 109
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 26 Gauge Quincke | 26 Gauge Atraucan | Total
Number analyzed (Participants) | 150 | 110 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 110 | 260
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.5) | 29.2 (4.8) | 29.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 110 | 260
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 150 | 110 | 260

OUTCOME MEASURES:

1. Primary Outcome: Postdural Puncture Headache in Patients Receiving Spinal Anesthesia for Cesarean Section
Description: Patients were observer for the symptoms of headache (PDPH) for 1 week. On the 1st postoperative day they were visited in the clinic. On the 7th postoperative day they were contacted by telephone and were asked about the symptoms.
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | 26 Gauge Quincke | 26 Gauge Atraucan
Number analyzed (Participants) | 147 | 109
participants | 14 | 10

2. Secondary Outcome: Backache in Patients Receiving Spinal Anesthesia for Cesarean Section
Description: Patients were observer for the symptoms of postdural puncture backache for 1 week. On the 1st postoperative day they were visited in the clinic. On the 7th postoperative day they were contacted by telephone and were asked about the symptoms.
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | 26 Gauge Quincke | 26 Gauge Atraucan
Number analyzed (Participants) | 147 | 109
participants | 65 | 68

ADVERSE EVENTS:
Time Frame: The patients were observed over one week period. No other extra observation was made as a routine. The stated adverse events had been reported during that time.
Description: One patient had sinus pause, that was observed just few minutes after the local anesthetic application. The second was found to have intracranial epidural hemathoma, that was found on the 1st postoperative day. We have linked it to minor head trauma 3 days before the surgery. The patient had not reported it in the anamnesis prior to the surgery.
Arm/Group | 26 Gauge Quincke | 26 Gauge Atraucan
Serious Adverse Events (participants affected / at risk) | 79/147 | 78/109
Other Adverse Events (participants affected / at risk) | 1/147 | 1/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 26 Gauge Quincke (N=147) | 26 Gauge Atraucan (N=109)
Postdural puncture headache (Nervous system disorders) | 14 (14) | 10 (10) — Postdural puncture headache (PDPH), a common side effect after spinal anesthesia. Can be serious.
Postdural puncture backache (Musculoskeletal and connective tissue disorders) | 65 (65) | 68 (68) — Postdural puncture backache (PDPB), a common side effect after spinal anesthesia. Rarely necessitates intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 26 Gauge Quincke (N=147) | 26 Gauge Atraucan (N=109)
Sinus rhythm pause (Cardiac disorders) | 0 (0) | 1 (1) — Sinus rhythm cessation for at least 3 seconds. Our patient had 6 second pause.
Epidural hemathoma (Nervous system disorders) | 1 (1) | 0 (0) — One patient had experienced intracranial epidural hemathoma. It was linked to the minor head trauma 3 days before the operation, which was missed out in the anamnesis.

LIMITATIONS AND CAVEATS:
We have planned to enroll 150 patients in the Atraucan group, but the circumstances forced us to finish the recruitment at 110.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No